CLINICAL TRIAL: NCT06626100
Title: SMART Family-Link Project: A Digital Game on Promoting Family Well-being
Brief Title: A Digital Game on Promoting Family Well-being
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Agnes Yuen-Kwan Lai, Principal Investigator, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW 20-353-2
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Family Research; Family-centered Care
Keywords: Gamification; Family well-being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise-themed game (Experimental): The intervention includes an exercise-themed quiz game and monitored step count.
  Interventions: Behavioral: Exercise-themed game
- Diet-themed game (Active Comparator): The intervention includes a diet-themed quiz game.
  Interventions: Behavioral: Diet-themed game

INTERVENTIONS:
Behavioral: Exercise-themed game — The intervention includes three parts: quiz questions on knowledge on and benefits of exercise; monitored step count using smartphone tracker; whatsapp reminders on the benefits of exercise.
  Arms: Exercise-themed game
Behavioral: Diet-themed game — The intervention includes two parts: quiz questions on knowledge on and benefits of healthy diet; whatsapp reminders on the benefits of healthy diet.
  Arms: Diet-themed game

SUMMARY:
Advances in information communication technologies (ICT) allow for ICT-assisted health promotion to become more common. Integrating ICT in health promotion has been suggested to offer many advantages compared to traditional approaches to promote family well-being. Research has also shown the positive effects of game-based approaches in enhancing health promotion interventions, especially with children. We will develop and conduct an online survey to assess the use of games and gamification for health promotion, as well as a family-based randomized controlled trial to promote healthy living.

DETAILED DESCRIPTION:
With growing emphasis on the development and maintenance of healthy lifestyles, the family role has increasing importance. A family-based health promotion strategy can be instrumental in helping disseminate and reinforce knowledge and behaviours on family well-being and better equip families to protect themselves and promote family well-being beyond the COVID-19 pandemic. Additionally, the pandemic led to increased sedentary behavior and unhealthy eating. New, innovative health promotion strategies and approaches to increase physical activity and healthy diet and enhance well-being are needed.

This study aims to investigate and use a game-based approach to enhance knowledge and behaviours on healthy living and family well-being. We will conduct quantitative and qualitative evaluation. The findings would provide evidence of the feasibility and effectiveness of such an approach in a family-based context. It would also guide the direction for future health education and awareness trials and related projects and campaigns for health promotion efforts and to help improve family well-being in the Hong Kong community and elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* Chinese-speaking;
* Parental consent for those under 18;
* Able to understand and play the game;
* Has a smartphone.

Exclusion Criteria:

• Individuals who cannot meet the inclusion criteria.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Step count | Baseline and one month
  Average daily step count

SECONDARY OUTCOMES:
Perceived improved family happiness | Baseline and one month
  Change assessed by a validated one-item Family Happiness scale (score from 0 to 10, higher scores indicate more family happiness).
Game satisfaction score | One month
  Overall game rating (on a scale of 0-5, higher scores indicate higher satisfaction).
Family well-being knowledge and behaviors | Baseline and one month
  Change assessed by outcome-based questions (scores from 0 to 10, higher scores indicate better knowledge and behaviors)
Self-reported healthy habits | Baseline and one month
  Change assessed by frequency-based questions related to exercise levels and consumption of fruits and vegetables (scores from 0 to 7 days, higher scores indicate more engagement in healthy habits)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Will share after the study is completed
Supporting Information: Study Protocol
Time Frame: After the study is completed
Access Criteria: The minimal anonymized dataset will be available upon request to interested researchers. For interested researchers, please contact, Ms Shirley Sit (email ssit@connect.hku.hk), (School of Public Health, The University of Hong Kong) for further information.

REFERENCES:
- [Background] Runacres A, Mackintosh KA, Knight RL, Sheeran L, Thatcher R, Shelley J, McNarry MA. Impact of the COVID-19 Pandemic on Sedentary Time and Behaviour in Children and Adults: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2021 Oct 27;18(21):11286. doi: 10.3390/ijerph182111286. PMID 34769800
- [Background] Ameryoun A, Sanaeinasab H, Saffari M, Koenig HG. Impact of Game-Based Health Promotion Programs on Body Mass Index in Overweight/Obese Children and Adolescents: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Child Obes. 2018 Feb/Mar;14(2):67-80. doi: 10.1089/chi.2017.0250. Epub 2017 Nov 29. PMID 29185787
- [Background] Chagas CMDS, Pontes E Silva TB, Reffatti LM, Botelho RBA, Toral N. Rango Cards, a digital game designed to promote a healthy diet: a randomized study protocol. BMC Public Health. 2018 Jul 24;18(1):910. doi: 10.1186/s12889-018-5848-0. PMID 30041639
- [Background] Edwards EA, Lumsden J, Rivas C, Steed L, Edwards LA, Thiyagarajan A, Sohanpal R, Caton H, Griffiths CJ, Munafo MR, Taylor S, Walton RT. Gamification for health promotion: systematic review of behaviour change techniques in smartphone apps. BMJ Open. 2016 Oct 4;6(10):e012447. doi: 10.1136/bmjopen-2016-012447. PMID 27707829